CLINICAL TRIAL: NCT07391891
Title: Use of Music Mindfulness for Pain Management in the ED Waiting Room
Brief Title: Musical Mindfulness for Pain in the ED Waiting Room
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Sean D Young, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00000311
Record Dates: First submitted 2025-11-18; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Music Therapy for Pain and Sedation; Neck Pain Musculoskeletal; Back Pain
Keywords: Music therapy; Music pain management; Musical pain managament; Opioid epidemic; Therapeutic medicine; Emergency Medicine; Emergency Room; Waiting Room; Music intervention; Jazz music; back pain; neck pain; musculoskeletal; musculoskeletal pain; pain; pain management; music
MeSH Terms: conditions — Back Pain; Emergencies; Neck Pain; Musculoskeletal Pain; Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients are blinded to condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Music Training + Music Intervention (Experimental): Participants will be given a video training on listening to music mindfully to reduce pain. Following this, patients will be given a 15-minute jazz music playlist to listen to.
  Interventions: Behavioral: Music intervention
- Standard of Care Pain Management Training + Participant's Choice of Intervention (Active Comparator): Participants will be given a video demonstrating how to mindfully manage pain, following this will be a 15-minute period of the participant's choice of activity
  Interventions: Behavioral: Music intervention

INTERVENTIONS:
Behavioral: Music intervention — Participant's will be taught how to mindfully listen to jazz to reduce pain

SUMMARY:
Studies have shown that 60-70% of patients in the Emergency Department (ED) experience pain. With pain being such a broad issue in the ED, the ED is expected to deliver safe and effective treatment of pain. However, with the current ongoing opioid epidemic, it is important to consider other methods, both pharmacologic and nonpharmacologic, of pain reduction. Jazz music specifically has been demonstrated to have therapeutic effects on pain that can be used to lower the quantity of opioids administered to patients.

Non-pharmacological interventions in the emergency department for pain typically consist of splinting an injury, applying heat or cold, or various distractions following initial and sequential pain assessment. Pharmacological interventions for pain in the Emergency Department involve the administration of acetaminophen, muscle relaxers, topical anesthetics, opioids, to name a few.

In the emergency department (ED), providers are increasingly hesitant to prescribe opioids over the past decade due to the current opioid epidemic, in which there is an increasing proportion of people that develop an addiction to opioids, including those that are prescribed to them for pain management.. While emergency medicine providers' decrease in opioid prescriptions pertains to their implementation of opioid-prescribing policies, little evidence has been found demonstrating a direct link in these policies to decreases in substance misuse. Consequently, providers find themselves needing to become ingenious in their approach to pain in patients through the integration of pharmacologic and non-pharmacologic mediums of analgesia.

A recent randomized controlled trial (RCT) from Brigham and Women's Hospital in Boston sought to identify the qualitative responses from patients in the ED following the arbitrary distribution of either supervised or unsupervised music therapy over a time period of 4 hours. The initial results found that, generally speaking, music therapy may lower reported pain and anxiety scores. Furthermore, stronger results were identified in case subjects with higher initial reports of pain via a pain catastrophizing scale, implying that a higher baseline of pain results in more relief from music therapy. One shortcoming in the article is the lack of analysis with reported results and the biopsychosocial model of pain. Heavy emphasis is placed on the psychological and social components of pain in the Brigham and Women's article through the implementation of the Pain Catastrophizing Scale and Brief Pain Inventory scoring done during the RCT, but no focus on linked biological changes in the subjects through the music therapy intervention.

The purpose of this study is to (i.) assess the effect of a video training about musical pain management followed by a 15-minute music listening intervention on self-reported pain scores in ED patients with neck and back pain. The investigators also aim to (ii.) evaluate patient satisfaction and emotional response following the intervention. Opioid medications are commonly used to reduce substantial pain, and music therapy has been found to reduce associated pain and anxiety in patients, then the use of music therapy could be an aid in medicine to reduce opioid intake. The investigators hypothesize that the usage of a training on musical pain management combined with a specified jazz musical intervention will produce a significantly lower measured pain score in comparison to a video on mindful pain management followed by the patient's choice of activities.

DETAILED DESCRIPTION:
1. Patients presenting to the Emergency Department with neck or back pain in the waiting room are approached for the study.
2. Researchers confirm patients' interest. Consent patient by having them sign the HIPAA Waiver and Informed Consent Form.
3. Obtain an initial pain measurement of the subject prior to randomization. Additionally, obtain demographic information about the subject
4. Randomize subjects into either the intervention group (mindful music listening video followed by jazz music playlist administration) or the control group (pain management video followed by video or music of participants choice administered) using a simple randomizer, such as the Sealed Envelope application.
5. Deliver musical pain management video (intervention group) OR allow for the current standard of care with pain management presentation video for 15 minutes (control group).
6. Deliver musical intervention to subjects in the intervention group for 15 minutes, or allow subjects in the control group to listen to music or video of their choice for 15 minutes.
7. Following the 15-minute music intervention or 15-minute control, obtain a new pain measurement
8. Follow up after 30 minutes after the music intervention finished and acquire pain measurements again
9. Follow up 1 hour after the music intervention finished and acquire pain measurements again
10. Administer brief survey to patient asking if they enjoyed or disliked the experience of the study and if they are likely or unlikely to participate again.

ELIGIBILITY:
Inclusion Criteria:

* - Age >= 18 years old and <=75 years old
* Patient presents with neck or back pain

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Pain score using Pain, Enjoyment of Life and General Activity Scale (PEG) | Day 1
  Pain score will be obtained using PEG scale
  Title of first scale: Pain Pain will be rated on a scale of 0-10 , with 0 being no pain, and 10 being pain as bad as you can imagine (pain increases as scale increases)
  Title of second scale: Interference Interference will be rated on a scale of 0-10, with 0 being no interference, and 10 being completely interferes (interference increases as scale increases) Higher score is a worse outcome
Pain Intensity | Day 1
  Pain will be scored using pain intensity scale Title of scale: Frequency 0-3, with 0 being not at all and 3 being nearly every day Higher score is a worse outcome

SECONDARY OUTCOMES:
Satisfaction with Study | 1 hour and 30 minutes after baseline
  Participants will be asked their satisfaction of the study to gauge if music therapy or mindful pain management is a feasible process in the Emergency Department Waiting Room
  How positive was your experience from 1-5, which 1 being horrible and 5 being amazing?
  How likely would you be to recommend this study to others undergoing similar pain, with 1 being not likely at all and 5 being extremely likely ?
  How easy was it to participate in this study from 1-5, with 1 being not easy at all, and 5 being extremely easy ?
  Would you consider undergoing this procedure again in the future? Yes or no, and why?

CONTACTS AND LOCATIONS:
Overall Officials: Sean Young, PhD, Principal Investigator — University of California, Irvine. Department of Emergency Medicine; Ryan Rokerya, Expected BS Dec 2026, Study Chair — University of California, Irvine. Department of Emergency Medicine; Tyler Mitchell, Expected BS Jun 2026, Study Chair — University of California, Irvine. Department of Emergency Medicine; Dominic A Ugarte, M.D., Study Chair — University of California, Irvine. Department of Emergency Medicine
Locations (1):
- University of California, Irvine, Emergency Department, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pourmand A, Jasani G, Shay C, Mazer-Amirshahi M. The Evolving Landscape of Acute Pain Management in the Era of the Opioid Crisis. Curr Pain Headache Rep. 2018 Aug 27;22(11):73. doi: 10.1007/s11916-018-0728-y. PMID 30151792
- [Background] Young SD, Kim J, Hanley A. Mindful Jazz and Preferred Music Interventions Reduce Pain Among Patients With Chronic Pain and Anxiety: A Pilot Randomized Controlled Trial. Cureus. 2025 Mar 12;17(3):e80485. doi: 10.7759/cureus.80485. eCollection 2025 Mar. PMID 40225443
- [Background] Chanana L, Jegaraj MA, Kalyaniwala K, Yadav B, Abilash K. Clinical profile of non-traumatic acute abdominal pain presenting to an adult emergency department. J Family Med Prim Care. 2015 Jul-Sep;4(3):422-5. doi: 10.4103/2249-4863.161344. PMID 26288785
- [Background] Chai PR, Schwartz E, Hasdianda MA, Azizoddin DR, Kikut A, Jambaulikar GD, Edwards RR, Boyer EW, Schreiber KL. A Brief Music App to Address Pain in the Emergency Department: Prospective Study. J Med Internet Res. 2020 May 20;22(5):e18537. doi: 10.2196/18537. PMID 32432550